CLINICAL TRIAL: NCT00693342
Title: A Randomized Phase III Trial in Patients With Epithelial Ovarian, Fallopian Tube or Peritoneal Cancer With a Polyvalent Vaccine-KLH Conjugate + OPT-821 Versus OPT-821
Brief Title: Vaccine Therapy and OPT-821 or OPT-821 Alone in Treating Patients With Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer in Complete Remission
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Never opened to accrual, a GOG working number, not developed into a clinical trial.
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000597674; GOG-OVM0703
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IA primary peritoneal cavity cancer; stage IB primary peritoneal cavity cancer; stage IC primary peritoneal cavity cancer; stage IIA primary peritoneal cavity cancer; stage IIB primary peritoneal cavity cancer; stage IIC primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; stage IV primary peritoneal cavity cancer; stage IA fallopian tube cancer; stage IB fallopian tube cancer; stage IC fallopian tube cancer; stage IIA fallopian tube cancer; stage IIB fallopian tube cancer; stage IIC fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

ARMS (2):
- Arm I (Experimental): Patients receive polyvalent antigen-KLH conjugate vaccine in combination with OPT-821 subcutaneously (SC) once in weeks 1, 2, 3, 7, 15, 27, 39, 51, 63, 75, and 87.
  Interventions: Biological: immunological adjuvant OPT-821; Biological: polyvalent antigen-KLH conjugate vaccine
- Arm II (Experimental): Patients receive OPT-821 SC once in weeks 1, 2, 3, 7, 15, 27, 39, 51, 63, 75, and 87.
  Interventions: Biological: immunological adjuvant OPT-821

INTERVENTIONS:
Biological: immunological adjuvant OPT-821 — Given subcutaneously
Biological: polyvalent antigen-KLH conjugate vaccine — Given subcutaneously
  Arms: Arm I

SUMMARY:
RATIONALE: Vaccines made from tumor antigens may help the body build an effective immune response to kill tumor cells. Biological therapies, such as OPT-821, may stimulate the immune system in different ways and stop tumor cells from growing. Giving vaccine therapy together with OPT-821 may kill more tumor cells. It is not yet known whether giving vaccine therapy together with OPT-821 is more effective than OPT-821 alone in treating ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

PURPOSE: This randomized phase III trial is studying vaccine therapy and OPT-821 to see how well they work compared with OPT-821 alone in treating patients with ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer in complete remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of patients with ovarian epithelial, fallopian tube, or primary peritoneal cancer in second or third complete clinical remission treated with a polyvalent antigen-KLH conjugate vaccine (GM2-KLH, Globo-H-KLH, Tn-MUC1-32mer-KLH, TF-KLH, and sTn-KLH) in combination with OPT-821 vs OPT-821 alone.

Secondary

* To compare the incidence of toxicities in patients treated with these regimens.
* To compare the overall survival of patients treated with these regimens.
* To characterize the immune response (by ELISA) in a limited sampling of patients, in order to determine if the outcome correlates with antigen-specific immune titers.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive polyvalent antigen-KLH conjugate vaccine in combination with OPT-821 subcutaneously (SC) once in weeks 1, 2, 3, 7, 15, 27, 39, 51, 63, 75, and 87.
* Arm II: Patients receive OPT-821 SC once in weeks 1, 2, 3, 7, 15, 27, 39, 51, 63, 75, and 87.

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for antibody expression to antigens (i.e., Tn-MUC1-32mer, GM2, Globo-H, TF, sTN, and Tn) by ELISA. IgM and IgG titers are also measured.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cancer

  * Any stage or grade at diagnosis allowed
* Has undergone initial cytoreductive surgery or received at least one platinum-based chemotherapy regimen

  * Recurred on initial therapy, but is now in second or third complete clinical remission as defined by the following:

    * Serum CA-125 normal
    * Negative physical examination
    * No definitive evidence of disease by CT scan of the abdomen and pelvis (lymph nodes and/or soft tissue abnormalities ≤ 1.0 cm are not considered definitive evidence of disease)

      * A positive PET scan is allowed provided other criteria are met and MRI or CT scan are negative
  * Completed last course of chemotherapy within the past 4 months

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2.0 times ULN
* SGOT ≤ 2.0 times ULN
* Alkaline phosphatase ≤ 2.0 times ULN

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Incidence of toxicities
Overall survival
Correlation of outcome with antigen-specific immune titers in a limited sampling of patients

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Jonathan S. Berek, MD — Stanford Comprehensive Cancer Center - Palo Alto